CLINICAL TRIAL: NCT07402551
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of RC1416 Injection in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Phase II Study of RC1416 Injection in COPD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing RegeneCore Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RJK-RC1416-301
Record Dates: First submitted 2026-01-28; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RC1416 Injection (Experimental)
  Interventions: Drug: RC1416
- Placebo Control (Placebo Comparator)
  Interventions: Drug: RC1416 Placebo

INTERVENTIONS:
Drug: RC1416 — There are two doses in this part. Each subjects will receive the drug by subcutaneous injection.
  Arms: RC1416 Injection
Drug: RC1416 Placebo — Each subjects will receive the placebo by subcutaneous injection.
  Arms: Placebo Control

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase II clinical study to evaluate the efficacy and safety of RC1416 injection in patients with moderate to severe chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Each participant will receive the study treatment once every two weeks for a total treatment duration of 52 weeks. The study aims to evaluate the annualized rate of moderate or severe COPD exacerbations (AECOPD) and the change in FEV1 from baseline over the 52-week treatment period. The changes in FeNO, total IgE, eosinophil count, and TARC levels from baseline will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 to 85 years (inclusive) at the time of signing the informed consent form, regardless of gender.
* Body Mass Index (BMI) ≥ 16 kg/m².
* Meets the diagnostic criteria for chronic obstructive pulmonary disease (COPD), and has medical records or relevant documentation indicating a history of COPD for ≥ 12 months at screening.
* Post-bronchodilator ratio of forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC) < 0.7, and post-bronchodilator FEV1 ≥ 30% and < 80% of the predicted value at screening.
* A current smoker or former smoker with a smoking history of ≥ 10 pack-years, or a history of exposure to other risk factors.
* A score of ≥ 2 on the modified Medical Research Council (mMRC) dyspnea scale at screening.
* Medical records or relevant documentation showing ≥ 2 moderate COPD. exacerbations (AECOPD) or ≥ 1 severe AECOPD within the 12 months prior to screening.
* Medical records or relevant documentation showing receipt of background triple therapy (ICS + LABA + LAMA) for ≥ 3 months prior to randomization.
* A blood eosinophil count ≥ 150/mm³ (0.15×10⁹/L) at screening.

Exclusion Criteria:

* A current diagnosis of asthma or a history of asthma.
* Presence of other significant pulmonary diseases except COPD as judged by the Investigator.
* History of malignancy .
* A history of autoimmune diseases , or treatment with biologics or systemic immunosuppressants for inflammatory diseases within 8 weeks or 5 half-lives (whichever is longer) prior to signing the informed consent form.
* Presence of recurrent, chronic, or other active infections at screening.
* Currently receiving or planning to start long-term oxygen therapy or mechanical ventilation during the study period.
* Diagnosis of α1-antitrypsin deficiency.
* Active hepatitis B, active hepatitis C, positive human immunodeficiency virus (HIV) antibody, or positive Treponema pallidum antibody (TP-Ab).
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-03-07 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
moderate or severe COPD exacerbations (AECOPD) and forced expiratory volume in 1 Second (FEV1) | During 52 weeks
  Evaluate the annualized rate of AECOPD and the change in FEV1 from baseline

SECONDARY OUTCOMES:
The safety and tolerability | During 52 weeks
  Adverse events, laboratory tests, vital signs, 12-lead electrocardiogram (ECG), and physical examinations.
pharmacokinetic | During 52 weeks
  Css, DF, Tmax.
immunogenicity | During 52 weeks
  ADA positivity rate and titer, and NAb positivity rate.
biomarkers predictive of the efficacy | During 52 weeks
  FeNO, total IgE, eosinophil count, and TARC levels.

CONTACTS AND LOCATIONS:
Locations (40):
- China (40):
  - Anhui Provincial Chest Hospital, Hefei, Anhui
  - Wan Bei General Hospital of Wanbei Coal power Group, Suzhou, Anhui
  - The Affiliated Bishan Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The first affiliated hospital of guangzhou medical university, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Huizhou Third People's Hospital, Huizhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Guangzhou Medical University Affiliated Qingyuan Hospital (Qingyuan People's Hospital), Qingyuan, Guangdong
  - The First Affiliated Hospital of guangxi Medical University, Nanning, Guangxi
  - The First People's Hospital of Yulin, Yulin, Guangxi
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Anyang People's Hospital, Anyang, Henan
  - Jiaozuo Second People's Hospital, Jiaozuo, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - Nanyang Second People's Hospital, Nanyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Xinxiang First People's Hospital, Xinxiang, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - Loudi Central Hospital, Loudi, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First People's Hospital of Lianyungang City, Lianyungang, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Yangzhou University Affiliated Hospital, Yangzhou, Jiangsu
  - Jiu Jiang NO.1 People's Hospital, Jiujiang, Jiangxi
  - People's Hospital of Pingxiang City, Pingxiang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - LiaoCheng People's Hospital, Liaocheng, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - The Second People's Hospital of Weifang, Weifang, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The Third People's Hospital of Chengdu City, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Mianyang central hospital, Mianyang, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Zigong First People's Hospital Zigong Academy of Medicalsciences, Zigong, Sichuan
  - The 2nd Affiliated Hospital and Yuying Children's Hospital of WMU, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No